CLINICAL TRIAL: NCT03891836
Title: Prevalence and Correlates of Depressive Symptoms Among Assiut University Medical Students
Brief Title: Depressive Symptoms Among Medical Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Medhat Soliman Gayed, Principle investigator, Assiut University
Other Study IDs: Students' depressive symptoms
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- medical students: All students from the chosen classes in each study year will be invited to complete self-administered questionnaire

SUMMARY:
Depression is a common mental disorder, people with depression feel sadness anxious, loss of interest or pleasure, hopeless, helpless, worthless feelings of guilt and poor concentration. It can impair person's ability to function at work or school, or cope with daily life. It can lead to suicide.

DETAILED DESCRIPTION:
Depressive symptoms are higher among women and its prevalence among university students was reported to be higher than the general population .There are various risk factors of depressive symptoms among university students, lower socioeconomic status, poor academic performance, overweight, life stressors, family history of psychiatric disorders, sleeping problems, and exposure to patients' suffering. Several studies were conducted among medical students in different Egyptian Universities to detect prevalence of depressive symptoms which were 42.9% in Al-Azhar Uni-versity, Cairo, 60.8% in Fayoum University, 59.2% in Mansoura University and 57.9% in Alexandria University.

A sense of control means having a feeling of autonomy, of choosing how you spend your time, of doing your own work in your own way, which is a key component of happiness. Depressive symptoms more common in those who feel there is little they can do to change important things in their lives.

Medical education is considered stressful. Medical students have psychological and academic stressors during their revolution from insecure students to young knowledgeable physicians, which were determined to be associated with depressive symptoms and decrease the quality of life and academic achievements.

ELIGIBILITY:
Inclusion Criteria:

All Egyptian medical students at faculty of Medicine, Assiut University in the academic year 2018-2019

Exclusion Criteria:

Non-Egyptian medical students

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian students registered at faculty of Medicine, Assiut University in the academic year 2018-2019
Sampling Method: Non-Probability Sample
Enrollment: 742 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of depressive symptoms among medical students by patient health questionnaire-9 | one year
  it is a scale used to diagnose major depressive disorder or other depressive disorder, each question in the scale take score from 0 to 3 summation of these scores detect degree of severity which is (1-4) minimal depression, (5-9) mild depression, (10-14) moderate depression, (15-19) moderately severe depression and (20-27) severe depression. It includes questions about: Lack of interest, depressed mood, sleeping difficulties, tiredness, appetite problems, negative feelings about self, concentration problems, psychomotor agitation/retardation and Suicidal ideation
social class of the student by family affluence sale III (FAS-III) | one year
  FAS consists of 6 items. The responses to the items are given as specific values and calculated as an aggregated FAS index ranging from 0 to 13. The more index of FAS-III the higher is social class of the student. It consists of questions about: motor vehicle, bedroom, computers, bathrooms, dishwasher and holidays.

SECONDARY OUTCOMES:
sense of control by MIDI scale | one year
  A sense of control means having a feeling of autonomy, of choosing how you spend your time, of doing your own work in your own way, which is a key component of happiness. Depressive symptoms more common in those who feel there is little they can do to change important things in their lives. This scale is a self-report measure of sense of control of 12 items. It measures sense of control in 2 categories:
  Perceived Constraints and Personal Mastery. The scores of 12 items will be averaged to create a composite measure. Higher scores indicated higher sense of control.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gayed, Principal Investigator — Assiut University
Locations (1):
- Assiut uiversity, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hope V, Henderson M. Medical student depression, anxiety and distress outside North America: a systematic review. Med Educ. 2014 Oct;48(10):963-79. doi: 10.1111/medu.12512. PMID 25200017
- [Background] Coentre R, Faravelli C, Figueira ML. Assessment of depression and suicidal behaviour among medical students in Portugal. Int J Med Educ. 2016 Oct 29;7:354-363. doi: 10.5116/ijme.57f8.c468. PMID 27794561
- [Background] Ibrahim AK, Kelly SJ, Glazebrook C. Socioeconomic status and the risk of depression among U.K. higher education students. Soc Psychiatry Psychiatr Epidemiol. 2013 Sep;48(9):1491-501. doi: 10.1007/s00127-013-0663-5. Epub 2013 Feb 15. PMID 23412652
- [Background] Ngin C, Pal K, Tuot S, Chhoun P, Yi R, Yi S. Social and behavioural factors associated with depressive symptoms among university students in Cambodia: a cross-sectional study. BMJ Open. 2018 Sep 28;8(9):e019918. doi: 10.1136/bmjopen-2017-019918. PMID 30269060
- [Background] Reyes-Rodriguez ML, Rivera-Medina CL, Camara-Fuentes L, Suarez-Torres A, Bernal G. Depression symptoms and stressful life events among college students in Puerto Rico. J Affect Disord. 2013 Mar 5;145(3):324-30. doi: 10.1016/j.jad.2012.08.010. Epub 2012 Aug 29. PMID 22939390
- [Background] Angelone AM, Mattei A, Sbarbati M, Di Orio F. Prevalence and correlates for self-reported sleep problems among nursing students. J Prev Med Hyg. 2011 Dec;52(4):201-8. PMID 22442926
- [Background] Bovero A, Tosi C, Miniotti M, Torta R, Leombruni P. Medical Students Reflections Toward End-of-Life: a Hospice Experience. J Cancer Educ. 2018 Jun;33(3):634-639. doi: 10.1007/s13187-017-1171-1. PMID 28130710
- [Background] Shams-Eldin AA, Hassan H, Abo Elkhar O et al. (2017): Prevalence of Depression among Medical Students at Al-Azhar Uni¬versity, Cairo, Egypt; Community Med Public Health: CMPH-115. DOI: 10.29011/CMPH-115/100015.
- [Background] Abdel Wahed W Y, Hassan S K. (2016): Prevalence and associated factors of stress, anxiety and depression among medical Fayoum University students; Alexandria Journal of Medicine Doi.org/10.1016/j.ajme.2016.01.005.
- [Background] Barakat D, Elwasify M et al. (2016): Relation between insomnia and stress, anxiety, and depression among Egyptian medical students; Middle East Current Psychiatry, Volume 23, Number 3, July 2016, pp. 119-127(9), DOI: https://doi.org/10.1097/01.XME.0000484345.57567.a9.
- [Background] Ibrahim MB, Abdelreheem MH. (2015): Prevalence of anxiety and depression among medical and pharmaceutical students in Alexandria/University Faculty of Medicine, Alexandria University. Alexandria J Med 2015;51:167-73.
- [Background] Wardle J, Steptoe A, Gulis G, Sartory G, Sek H, Todorova I, Vogele C, Ziarko M. Depression, perceived control, and life satisfaction in university students from Central-Eastern and Western Europe. Int J Behav Med. 2004;11(1):27-36. doi: 10.1207/s15327558ijbm1101_4. PMID 15194517
- [Background] Alzahrani AHS. (2017): Depression and suicide among medical students: a comparison study between medical and medical sciences students in Taif University, Taif-KSA. W J Pmr., 3(2):1822.
- [Background] Pillay N, Ramlall S, Burns JK. Spirituality, depression and quality of life in medical students in KwaZulu-Natal. S Afr J Psychiatr. 2016 Mar 22;22(1):731. doi: 10.4102/sajpsychiatry.v22i1.731. eCollection 2016. PMID 30263152